CLINICAL TRIAL: NCT01241825
Title: The Effect of Chewing Gum on Small Bowel Transit Time: a Prospective Randomized Trial.
Brief Title: The Effect of Chewing Gum on Small Bowel Transit Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H10-01726
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Bowel Transit Times
Keywords: capsule endoscopy; chewing gum; small bowel transit time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Active Comparator): The subject group will chew sugarless chewing gum for a specific amount of time while undergoing capsule endoscopy.
  Interventions: Other: Trident sugarless chewing gum.
- 2. (Placebo Comparator): The control group will not chew chewing gum while undergoing capsule endoscopy.
  Interventions: Other: One control group (these do not chew gum).

INTERVENTIONS:
Other: Trident sugarless chewing gum. — Patients will be randomly divided into 2 groups, one subject group (these chew gum) and one control group (these do not chew gum). The subjects will have to chew Trident sugarless chewing gum for 20-30 minutes every 2 hours, all together 4 times at t=0 h, t=2, t=4 and t=6 h.
  Arms: 1.
Other: One control group (these do not chew gum). — The control group will not chew chewing gum while undergoing capsule endoscopy
  Arms: 2.

SUMMARY:
The purpose of this study is to see if chewing sugarless chewing gum alters the time it takes for a capsule endoscopy to travel through the stomach and small bowel, and to see if more/less capsule endoscopes reach the large bowel.

DETAILED DESCRIPTION:
The subjects will include patients already referred to us for a capsule endoscopy (CE) in this unit. We have calculated how many patients we need from small bowel transit times from the last 100 patients who had a CE at our centre. We will include 122. These will be randomly divided into two groups. The patients (chew chewing gum) and the controls (do not chew chewing gum).

ELIGIBILITY:
Inclusion Criteria:

* All out-patients > 19 years old presenting for capsule endoscopy

Exclusion Criteria:

* Patients on narcotics
* Patients on motility enhancing and/or slowing drugs should stop these at least 5 days prior to the procedure or be excluded from the study.
* Patients, who have proven or suspected obstruction of the bowel.
* Patients, who have had prior small bowel and/or gastric surgery.
* Patients with an ileostomy.
* Patients who have a known and/or have a history of swallowing disorder
* Patients with diabetes and/or hypo-/hyper- thyroidism
* Patients in whom the capsule become impacted at a stricture (these patients will be taken out of the study and given the necessary medical/surgical treatment).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Small bowel transit time | 6 hours

SECONDARY OUTCOMES:
Gastric transit time, cecal completion rate | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Enns, Dr., Principal Investigator — University of British Columbia; Eric Lam, Dr., Study Director — University of British Columbia; Jennifer Telford, Dr., Study Director — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ou G, Svarta S, Chan C, Galorport C, Qian H, Enns R. The effect of chewing gum on small-bowel transit time in capsule endoscopy: a prospective, randomized trial. Gastrointest Endosc. 2014 Apr;79(4):630-6. doi: 10.1016/j.gie.2013.08.038. Epub 2013 Oct 7. PMID 24112594